CLINICAL TRIAL: NCT02029976
Title: School Nurse-directed Secondary Obesity Prevention for Elementary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00029947; 1R01NR013473-01A1 (NIH)
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- attention control condition (Active Comparator): Child and parent participants randomized to the attention control condition will receive a Newsletter Program or mailed monthly newsletter with general family-focused health information.
  Interventions: Behavioral: Mailed monthly newsletters
- after school weight management program (Experimental): The 9-month after school weight management program called SNAPSHOT (Student, Nurses and Parents Seeking Healthy Options Together), with a focus on healthy food and activity practices will be directed by a school nurse and will include: 1) quarterly parent/child coaching sessions with the school nurse held in the participant's home; 2) 14 child group sessions led by the school nurse, held in a school setting 1-2 times a month; 3) 5 parent group sessions led by a school nurse held in a school setting.
  Interventions: Behavioral: SNAPSHOT (Student, Nurses and Parents Seeking Healthy Options Together)

INTERVENTIONS:
Behavioral: SNAPSHOT (Student, Nurses and Parents Seeking Healthy Options Together) — attention control condition after school weight management program
  Arms: after school weight management program
Behavioral: Mailed monthly newsletters — Newsletters
  Arms: attention control condition

SUMMARY:
Primary Aim: To test the efficacy of an elementary school-based, school nurse-led weight management program to reduce excess weight gain among children, 8 to 12 years old who are overweight and at risk of overweight by increasing healthy dietary practices and physical activity levels and decreasing sedentary practices.

Primary Hypothesis: Relative to the control condition, the children receiving the intervention will have a significantly lower body mass index (BMI), following implementation of the 9-month intervention, controlling for baseline values.

DETAILED DESCRIPTION:
Primary Hypothesis: Relative to the control condition, the children receiving the intervention will have a significantly lower body mass index (BMI), following implementation of the 9-month intervention, controlling for baseline values.

ELIGIBILITY:
Inclusion Criteria for child participants:

* 3rd 4th and 5th grade student the year the intervention is implemented,
* ≥ 8 and ≤ 12 years old,
* age- and gender-adjusted BMI ≥ 75th percentile,
* child must live in a primary residence with the participating parent

Exclusion Criteria for child participants:

* plans to move outside the school district within the next 12 months,
* food allergies,
* physical limitations,
* medical conditions that prohibit participation in the intervention program or measurement,
* does not speak and write in English.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Actual)
Dates: Start 2014-04; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Kubik, PhD, Principal Investigator — Temple University
Locations (3):
- United States (3):
  - University of Massachusetts Amherst, Amherst, Massachusetts
  - University of Minnesota School of Nursing, Minneapolis, Minnesota
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kubik MY, Gurvich OV, Fulkerson JA. Association Between Parent Television-Viewing Practices and Setting Rules to Limit the Television-Viewing Time of Their 8- to 12-Year-Old Children, Minnesota, 2011-2015. Prev Chronic Dis. 2017 Jan 19;14:E06. doi: 10.5888/pcd14.160235. PMID 28103183
- [Background] Schroeder K, Kubik MY, Lee J, Sirard JR, Fulkerson JA. Self-Efficacy, Not Peer or Parent Support, Is Associated With More Physical Activity and Less Sedentary Time Among 8- to 12-Year-Old Youth With Elevated Body Mass Index. J Phys Act Health. 2020 Jan 1;17(1):74-79. doi: 10.1123/jpah.2019-0108. PMID 31756720
- [Background] Lee J, Kubik MY, Fulkerson JA. Missed Work Among Caregivers of Children With a High Body Mass Index: Child, Parent, and Household Characteristics. J Sch Nurs. 2021 Oct;37(5):396-403. doi: 10.1177/1059840519875506. Epub 2019 Sep 12. PMID 31514567
- [Background] Lee J, Kubik MY, Fulkerson JA. Diet Quality and Fruit, Vegetable, and Sugar-Sweetened Beverage Consumption by Household Food Insecurity among 8- to 12-Year-Old Children during Summer Months. J Acad Nutr Diet. 2019 Oct;119(10):1695-1702. doi: 10.1016/j.jand.2019.03.004. Epub 2019 May 2. PMID 31056369
- [Background] Kubik MY, Fulkerson JA, Sirard JR, Garwick A, Temple J, Gurvich O, Lee J, Dudovitz B. School-based secondary prevention of overweight and obesity among 8- to 12-year old children: Design and sample characteristics of the SNAPSHOT trial. Contemp Clin Trials. 2018 Dec;75:9-18. doi: 10.1016/j.cct.2018.10.011. Epub 2018 Oct 18. PMID 30342255
- [Background] Dozier SGH, Schroeder K, Lee J, Fulkerson JA, Kubik MY. The Association between Parents and Children Meeting Physical Activity Guidelines. J Pediatr Nurs. 2020 May-Jun;52:70-75. doi: 10.1016/j.pedn.2020.03.007. Epub 2020 Mar 19. PMID 32200320
- [Background] Lee J, Kubik MY, Fulkerson JA. Media Devices in Parents' and Children's Bedrooms and Children's Media Use. Am J Health Behav. 2018 Jan 1;42(1):135-143. doi: 10.5993/AJHB.42.1.13. PMID 29320346
- [Derived] Lee J, Helgeson E, Horning ML, Elgesma KM, Kubik MY, Fulkerson JA. Food Insecurity and Changes in Diet Quality and Body Mass Index z-Scores Among Elementary School Students. Child Obes. 2024 Oct;20(7):508-516. doi: 10.1089/chi.2023.0185. Epub 2024 Mar 28. PMID 38546529
- [Derived] Kubik MY, Lee J, Fulkerson JA, Gurvich OV, Sirard JR. School-Based Secondary Obesity Prevention for Eight- to Twelve-Year-Olds: Results from the Students, Nurses, and Parents Seeking Healthy Options Together Randomized Trial. Child Obes. 2021 Apr;17(3):185-195. doi: 10.1089/chi.2020.0321. Epub 2021 Feb 18. PMID 33601934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohorts of children along with a parent were recruited annually from 2014 to 2017 and January through May, for a total of 4 cohorts. Data analyses of primary and secondary outcomes did not occur until cohort 4 completed the year 2: follow up measurement in August 2019.
Groups:
- After School Weight Management Program: The 9-month after school weight management program called SNAPSHOT (Student, Nurses and Parents Seeking Healthy Options Together), with a focus on healthy food and activity practices will be directed by a school nurse and will include: 1) quarterly parent/child coaching sessions with the school nurse held in the participant's home; 2) 14 child group sessions led by the school nurse, held in a school setting 1-2 times a month; 3) 5 parent group sessions led by a school nurse held in a school setting;
Period: YR-1 Post Intervention vs Baseline
Arm/Group | Attention Control Condition | After School Weight Management Program
Started | 132 | 132
Completed | 120 | 124
Not Completed | 12 | 8
Not completed — Lost to Follow-up | 12 | 8
Period: YR-2 Follow Up vs Baseline
Arm/Group | Attention Control Condition | After School Weight Management Program
Started | 132 (Attrition at end of year 2 was calculated based on baseline enrollment) | 132 (Attrition at end of year 2 was calculated based on baseline enrollment)
Completed | 122 | 124
Not Completed | 10 | 8
Not completed — Lost to Follow-up | 8 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Moved from area | 0 | 2

BASELINE CHARACTERISTICS:
Population: Per condition, at baseline, there were 66 child participants and 66 adult/parent participants .
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control Condition | After School Weight Management Program | Total
Number analyzed (Participants) | 132 | 132 | 264
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 66 | 66 | 132
  Between 18 and 65 years | 66 | 66 | 132
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per condition, at baseline, there were 66 child participants and 66 adult/parent participants, totaling 132 per condition and 264 overall
  years
    Child participants: number analyzed (Participants) | 66 | 66 | 132
    Child participants | 9.3 (0.9) | 9.3 (0.9) | 9.3 (0.9)
    Adult/parent participants: number analyzed (Participants) | 66 | 66 | 132
    Adult/parent participants | 38.9 (6.7) | 39.3 (7.4) | 39.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Per condition, at baseline, there were 66 child participants and 66 adult/parent participants, totaling 132 per condition and 264 overall
  Participants
    Child participants: number analyzed (Participants) | 66 | 66 | 132
    Child participants: Female | 31 | 34 | 65
    Child participants: Male | 35 | 32 | 67
    Adult/parent participants: number analyzed (Participants) | 66 | 66 | 132
    Adult/parent participants: Female | 61 | 63 | 124
    Adult/parent participants: Male | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Per condition, at baseline, there were 66 child participants and 66 adult/parent participants, totaling 132 per condition and 264 overall
  Participants
    Child participants: number analyzed (Participants) | 66 | 66 | 132
    Child participants: White | 25 | 24 | 49
    Child participants: Hispanic | 15 | 15 | 30
    Child participants: Black | 15 | 13 | 28
    Child participants: Other | 11 | 14 | 25
    Adult/parent participants: number analyzed (Participants) | 66 | 66 | 132
    Adult/parent participants: White | 36 | 40 | 76
    Adult/parent participants: Hispanic | 14 | 12 | 26
    Adult/parent participants: Black | 8 | 9 | 17
    Adult/parent participants: Other | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 132 | 132 | 264
BMIz [Mean (Standard Deviation); unit: units on a scale] — Population: Value of the primary outcome, child BMIz, at baseline.
  units on a scale
    number analyzed (Participants) | 66 | 66 | 132
    (all) | 1.7 (0.7) | 1.5 (0.6) | 1.6 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Child Body Mass Index (BMI)
Description: Body Mass Index (primary outcome) is the recommended method of assessing overweight among children and was calculated with the formula: weight (kg)/height (m) 2. To determine child BMI percentile, we calculated age- and gender-adjusted BMI with Centers for Disease Control and Prevention (CDC) growth charts.. The primary outcome measure is BMI Z-Score, which indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. A higher Z-score is a less favorable outcome when assessing overweight/obesity across conditions in a healthy weight management intervention..
Time Frame: Measurement data will be collected at baseline prior to randomization and 12 (YR-1 post intervention), and 24 (YR-2 follow up) months post randomization
Population: Analysis population for primary outcome of BMI Z-score was child participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Control Condition | After School Weight Management Program
Number analyzed (Participants) | 61 | 62
units on a scale
  YR-1 Post Intervention: number analyzed (Participants) | 60 | 62
  YR-1 Post Intervention | 1.6 (0.7) | 1.5 (0.7)
  YR-2 Follow Up | 1.7 (0.7) | 1.6 (0.6)

2. Secondary Outcome: Dietary: Healthy Eating Index
Description: The Healthy Eating Index-2015 (HEI-2015) will be assessed with multiple 24-hour dietary recall interviews. A score on the HEI-2015 ranges from 0 to 100, with 100 meeting the recommendations for all 13 components of the HEI-2015. The higher the score the better.
Time Frame: The measure was collected at 12 months (YR-1 post intervention) following randomization with result adjusted for baseline value, percent body fat, sex and economic assistance
Population: Child participants who completed 24-hour dietary recall at baseline and 12-months post randomization, following completion of the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Control Condition | After School Weight Management Program
Number analyzed (Participants) | 55 | 55
units on a scale | 47.6 (12.5) | 51.9 (13.0)

3. Secondary Outcome: Activity
Description: Activity will be assessed with the MTI ActiGraph uniaxial accelerometer worn for a 7-day period. Time spent in each category of sedentary or moderate-vigorous physical activity was calculated as a percent of total wear time, with higher numbers indicating more time spent in the category.
Time Frame: The measure was collected at 12 months (YR-1 post intervention), following randomization with result adjusted for baseline value, percent body fat, sex and age
Population: Child participants were required to provide at least 480-minutes of wear time per day to represent a day of data. Participants with 2-3 days of wear time underwent a within-participant "imputation" method that used all available data to create a composite day.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Attention Control Condition | After School Weight Management Program
Number analyzed (Participants) | 51 | 50
percentage of time
  Moderate or Vigorous Physical Activity (MVPA) | 4.5 (2.7) | 4.2 (2.9)
  Sedentary Behavior | 67.2 (8.5) | 67.6 (8.2)

4. Secondary Outcome: Total Quality of Life
Description: The 23-item Pediatric Quality of Life (QOL) child inventory or PedsQL 4.0 was used to assess physical, emotional, social and school functioning. Responses are reversed scored and transformed to a 0 to 100 scale which is used to calculate a total health-related quality of life summary score (mean of 23 items) which includes a physical health summary score (mean of 8 physical functioning items) and psycho-social health summary score (mean of 15 emotional, social and school functioning items). A higher score indicates better child-reported health-related quality of life.
Time Frame: Measurement data will be collected at baseline prior to randomization and 12 (YR-1 post intervention) , and 24 (YR-2 follow up) months following randomization
Population: analysis population included children who provided survey data at baseline and 12- and 24-months post randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Control Condition | After School Weight Management Program
Number analyzed (Participants) | 61 | 62
units on a scale
  Year One Post Intervention | 76.0 (16.3) | 72.3 (16.1)
  Year Two Follow Up | 78.3 (14.7) | 77.0 (15.4)

ADVERSE EVENTS:
Time Frame: Monitoring for adverse events occurred for each participant from baseline data collection to completion of follow up measurement and encompassed measurement and intervention activities.
Description: Definitions as per clinicaltrials.gov
Arm/Group | Attention Control Condition | After School Weight Management Program
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/132
Other Adverse Events (participants affected / at risk) | 0/132 | 0/132

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT02029976/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT02029976/SAP_001.pdf